CLINICAL TRIAL: NCT03558321
Title: Relation Between Human Epididymis Protein 4 (HE4) and Endometrial Pathology in Patients With Postmenopausal Bleeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Maged, professor, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 37
Record Dates: First submitted 2018-06-04; First posted 2018-06-15 (Actual); Last update posted 2018-06-15 (Actual); Status verified 2018-06

CONDITIONS: Postmenopausal Bleeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- post menopausal bleeding (Experimental): women with postmenopausal bleeding and endometrial thickness more than 5 mm
  Interventions: Procedure: Hysteroscopic guided fractional curretage; Procedure: total abdominal hysterectomy, bilateral salpingo oophrectomy, with or without pelvic lymph nodal dissection

INTERVENTIONS:
Procedure: Hysteroscopic guided fractional curretage — Under general anaesthesia , evaluation of the endometrial cavity was done followed by biopsy of the whole endometrial tissue
Procedure: total abdominal hysterectomy, bilateral salpingo oophrectomy, with or without pelvic lymph nodal dissection — Through abdominal incision , removal of the whole uterus , both tubes and ovaries and in some cases pelvic lymph nodes removal was done

SUMMARY:
All patients included in the study had single or multiple episodes of postmenopausal bleeding with an endometrial thickness of more than 5mm.

full history, general and local examination were done. Transvaginal ultrasound (TVS) was performed .The uterus was scanned in the sagittal plane. The double-layer ET was measured at the widest point between the endometrial-myometrial interfaces.the level of HE4 was measured. All women underwent hystrospopic guided endometrial biopsy. Definitive management was later performed in the form of total abdominal hysterectomy, bilateral salpingo oophrectomy, with or without pelvic lymph nodal dissection and histopathological examination.

DETAILED DESCRIPTION:
All patients included in the study had single or multiple episodes of postmenopausal bleeding with an endometrial thickness of more than 5mm.

Full history was taken , the number of episodes of postmenopausal bleeding, and previous investigations and current medications), general examination was performed and local examination was performed for all patients.

Transvaginal ultrasound (TVS) was performed .The uterus was scanned in the sagittal plane. The double-layer ET was measured at the widest point between the endometrial-myometrial interfaces by using electronic calipers. If there was fluid in the uterine cavity it was recorded. Suspected polyp was also recorded.

For the level of HE4: 5 ml of venous blood were withdrawn from all patients. The samples were left to clot. The separated sera were stored at -20˚ until all samples were obtained. Frozen samples were allowed to reach room temperature prior to use. Samples were then mixed thoroughly by gently inverting multiple times before analysis. HE4 was quantitatively assayed using the enzyme immunoassay (EIA) method (Fujirebio Diagnostics, Inc. Göteborg, Sweden). The functional sensitivity of the HE4 EIA is ≤ 25pM. The analytical specificity is 100 ± 15%.

All patients were then submitted to hysteroscopy under general anesthesia and endometrial biopsy.

After hysteroscopy and biopsy, 2 patient proved to have cervical malignancy, 2 patients were unfit for open surgery, and another 6 patients did not show up after. These 10 patients were excluded from the study leaving 90 patients eligible for final analysis .

Definitive management was later performed in the form of total abdominal hysterectomy, bilateral salpingo oophrectomy, with or without pelvic lymph nodal dissection and histopathological examination.

ELIGIBILITY:
Inclusion Criteria:

* Patients with single or multiple episodes of postmenopausal bleeding Endometrial Thickness ≥ 5mm

Exclusion Criteria:

* • History of other Malignancies

  * Patients on chemo and/or radiotherapy
  * Patients on tamoxifen
  * Patients unfit for surgical intervention
  * Patients on HRT or other hormonal treatment

Ages: 50 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 100 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
endometrial pathology | 3 days after hystroscopy
  pathological examination of the endometrial tissue

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, Principal Investigator — professor
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided